CLINICAL TRIAL: NCT01207193
Title: Effect of Bone Marrow-derived Mesenchymal Stem Cell Transplantation in Reconstructing Bone Defects.
Brief Title: Treatment Of Bone Cyst With Bone Marrow Mesenchymal Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Hamid Gourabi/President of Royan Institute, Royan Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Bone-005
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2009-03

CONDITIONS: Bone Cyst
Keywords: bone cyst bone defect mesenchymal cell
MeSH Terms: conditions — Bone Cysts | interventions — Carboxylesterase; Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bone cyst (Experimental): Patients with bone cyst defect are injected with mesenchymal cells.
  Interventions: Biological: cell injection

INTERVENTIONS:
Biological: cell injection — injection of mesenchymal cells to bone cyst defect
  Other Names: cell transplantation

SUMMARY:
There are two types of bone cysts, unicameral and aneurismal. These cysts happen to anyone, but they are most commonly seen in children and young adults while their bones are still growing. Living with a bone cyst and determining treatment options depend on the type of cyst.

Non-surgical treatments for unicameral bone cysts involves repeated X-rays in individuals who do not experience any symptoms.

Surgical removal of a unicameral bone cyst is needed if it becomes especially painful, or the area of the bone starts to thin out. The investigators aim to assess the clinical efficacy and side effects of mesenchymal stem cells seeded on bone matrix in repairing bone cyst.

DETAILED DESCRIPTION:
Bone cysts are benign lesions usually discovered in children from age of 5 to 15 years. Treatment options include observation, corticosteroid injection and surgery. Sometimes the risk of surgery is comparable to the likelihood of fracture without treatment. In orthopedic surgery, bone chips , various types of ceramics, natural and synthetized bone mineral hydroxyapatite and tricalcium phosphate, as well as numerous polymers and co-polymers of alfa-hydroxy acids are used to perform as an osteoconductive and rarely osteoinductive factor to help bone formation.Some evidence demonstrated that bone marrow mesenchymal stem cells deposited on the surface of this constructs enhance its osteogenic differentiation. In this study the investigators seeds cultured bone marrow derived mesenchymal stem cells on bone matrix, to evaluate its therapeutic potential in repairing unicameral or aneurysmal bone cyst.This composite is placed in the bone cyst after its curettage during a surgery.Post-operation assessment is done by X-Ray examination and MRI at 1, 2, 6, and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Bone cyst diagnosed with MRI, CT-scan, or X-Ray
* Intact cyst wall with high risk for fracture
* Cysts with minimum diameter of 6mm
* Diagnostic test performed on cyst fluid
* Provided written consent form

Exclusion Criteria:

* Patients with diagnosis of cancer
* Patients enrolled in other clinical trial

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
fulfill bone cyst defect | 6 months
  Defect of bone due to cyst fulfill after cell transplantation.

SECONDARY OUTCOMES:
effect of mesenchymal cell transplantation | 6 months
  Evaluate effect of mesenchymal cell transplantation to fulfill the defect of bone cyst.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — President of Royan Institute; Mohammad reza Baghban Eslami Nejad, PhD, Study Director — Scientific Board; Mohssen Emadeddin, MD, Principal Investigator — Orthopedic Investigator; Ahmad Vosough, MD, Study Director — Radiologist investigator; Nasser Aghdami, MD,PhD, Principal Investigator — Head of regenerativ center
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Royan Institute — http://www.royaninstitute.org